CLINICAL TRIAL: NCT00564083
Title: Randomized Controlled Trial Comparing Acellular Collagen Biomesh (Pelvisoft) to Polypropylene Mesh(Pelvitex) for Sacral Colpopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Health System (Other)
Responsible Party: Patrick Culligan MD, Atlantic Health System
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: BARD
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2007-11

CONDITIONS: Uterine Prolapse
Keywords: Compare the relative differences between the organic and sythentic materials for sacryl colpopexy.
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: sacral colpopexy — This surgery involves supporting the prolapsed vaginal wall with a piece of material (known as a graft) attached to a ligament along your backbone (or sacrum)

SUMMARY:
This research protocol is a randomized controlled trial. It is being done to compare and find out the relative differences between the materials, (Pelivisoft) "natural organic mesh" to poly propylene mesh (Pelvitex) "manmade mesh" after a surgery known as sacral colpopexy. This surgery involves supporting the prolapsed vaginal wall with a piece of material (known as a graft) attached to a ligament along your backbone (or sacrum). These materials are both FDA approved and widely used. The following objectives: anatomic outcomes, graft-related complications between the two materials, changes in pelvic organ prolapse-related quality of life, subjective changes in sexual function,changes in bowel function and the prolapse related pain present after sacral colpopexy will be evaluated.

The study visits are all under standard of care. Study questionnaires are unique to the study and will be completed at the enrollment in hospital, 2, 6,12 weeks, 6 months and one year visits The questionnaires are related to bowel function, bladder function, prolapse and sexual activity.

Permission will be requested to contact the patient again 5 years after surgery. Contact in the future will in no way obligate the patient to participate.

There may or may not be direct medical benefits to the participant. Decreased risk of erosion may be a possible benefit if placed in the organic "natural" arm of the study. The information learned from this study may benefit other patients in the future

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age

Exclusion Criteria:

* Prior sacral colpopexy or rectopexy

Contraindication to surgery based on co-existent medical condition

Desire for expectant management or pessary use

Pregnancy or the desire for pregnancy within 24 months of the sacral colpopexy procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-12; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
anatomic outcomes,graft-related complications between the two materials, changes in pelvic organ prolapse-related quality of life,subjective changes in sexual function,changes in bowel function and the prolapse related pain present after sacral colpopexy | One year

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Culligan, MD, Principal Investigator — Atlantic Health Urogynecology
Locations (1):
- Urogynecology, 95 Madison Ave., Morristown, New Jersey, United States

REFERENCES:
- [Derived] Culligan PJ, Salamon C, Priestley JL, Shariati A. Porcine dermis compared with polypropylene mesh for laparoscopic sacrocolpopexy: a randomized controlled trial. Obstet Gynecol. 2013 Jan;121(1):143-51. doi: 10.1097/aog.0b013e31827558dc. PMID 23262939